CLINICAL TRIAL: NCT06522165
Title: Pediatric Oncological Orthopaedic Reconstruction : "Analysis of the Clinical and Radiographic Results"
Brief Title: Pediatric Oncological Orthopaedic Reconstruction
Status: Active, not recruiting | Type: Observational
Sponsor: Costantino Errani (Other)
Responsible Party: Sponsor-Investigator, Costantino Errani, Principal Investigator, Istituto Ortopedico Rizzoli
Organization: Istituto Ortopedico Rizzoli (Other)
Other Study IDs: ROP
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Bone Tumor; Bone Cancer
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients: Male and female patients surgically treated with an oncological reconstructions at Rizzoli Orthopaedic Institute between 01/01/1991 and 31/12/2023
  Interventions: Other: Analysis

INTERVENTIONS:
Other: Analysis — analysis and review of imaging and clinical data

SUMMARY:
From the archives of the Rizzoli institute all the children undergoing oncological reconstruction from 1991 to 2023 (approximately 400 patients). A review will be made of the medical records, radiological imaging, and histological data of these patients

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bone sarcoma
* Patients with available clinical and imaging data

Exclusion Criteria:

* At least one inclusion criteria not met

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Male and female pediatric patients surgically treated with an oncological reconstruction from 1991 to 2023
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
longevity of the reconstruction | at baseline (day 0)
  -assess the longevity associated with pediatric oncologic reconstructions;

SECONDARY OUTCOMES:
complications | at baseline (day 0)
  assess the complications associated with pediatric oncologic reconstructions;

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Itituto Ortopedico Rizzoli, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abdeen A, Hoang BH, Athanasian EA, Morris CD, Boland PJ, Healey JH. Allograft-prosthesis composite reconstruction of the proximal part of the humerus: functional outcome and survivorship. J Bone Joint Surg Am. 2009 Oct;91(10):2406-15. doi: 10.2106/JBJS.H.00815. PMID 19797576
- [Background] Aponte-Tinao LA, Ayerza MA, Muscolo DL, Farfalli GL. Allograft reconstruction for the treatment of musculoskeletal tumors of the upper extremity. Sarcoma. 2013;2013:925413. doi: 10.1155/2013/925413. Epub 2013 Feb 14. PMID 23476115
- [Background] Azoury SC, Shammas RL, Othman S, Sergesketter A, Brigman BE, Nguyen JC, Arkader A, Weber KL, Erdmann D, Levin LS, Kovach SJ, Innocenti M. Outcomes following Free Fibula Physeal Transfer for Pediatric Proximal Humerus Reconstruction: An International Multi-Institutional Study. Plast Reconstr Surg. 2023 Apr 1;151(4):805-813. doi: 10.1097/PRS.0000000000010001. Epub 2022 Dec 6. PMID 36729876